CLINICAL TRIAL: NCT00941850
Title: TRIple-site VENTricular Pacing in Non-responders to Conventional Dual Ventricular Site Cardiac Resynchronization Therapy
Brief Title: A Study of Triple-site Ventricular Pacing in Patients Who Have Not Responded to Conventional Dual Ventricular Site Cardiac Resynchronization Therapy
Acronym: TRIVENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHL10707
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronizton therapy; CRT; Heart failure; Dyssynchrony; Echocardiography; Pacemakers; Nonresponders
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Triple site CRT (Experimental): These patients will continue to receive CRT via existing device but will have a change in the mode of delivery of therapy (by placing a second pacing lead to reach a different part of the left ventricle from the part originally paced
  Interventions: Procedure: Upgrade to triple ventricular site CRT
- Optimised medical and device therapy (No Intervention): These patients will receive optimised medical and device therapy.

INTERVENTIONS:
Procedure: Upgrade to triple ventricular site CRT — Patients in this arm will continue to receive CRT via the original unit, but some will have a change in the mode of delivery of therapy (by placing a second pacing lead to reach a different part of the left ventricle from the part originally paced).
  Arms: Triple site CRT

SUMMARY:
Patients are randomised to receive ongoing optimised device and medical therapy or triple ventricular site resynchronisation. The hypothesis states that patients receiving triple-site resynchronization will exhibit a better response.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a CRT device > 6 months previously according to current and conventional CRT indications
* Device optimization > 1 months previously
* Aged 18yrs or older
* Able to attend outpatient follow up

Exclusion Criteria:

* Recent MI (<2 months)
* Women who are pregnant or planning pregnancy
* Severe co morbid illness (where patients are not expected to survive duration of follow up period or where repeated outpatient visits may not be in best interest of patients)
* Upgrade procedure is contraindicated for safety reasons.
* Class IV inotropic agents
* Patient unwilling to comply with required follow-up protocol including randomization scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Proportion of responders in each group. o Clinical response will be defined according to the Packer score o Echocardiographic response will be defined as a 10% relative reduction in left ventricular end systolic volume at six months | 6 months

SECONDARY OUTCOMES:
NYHA class | 3 and 6 months
ECHO parameters (LVEDV/ESV, LVEF, MR severity, dyssynchrony indices: time to peak velocity/strain/deformation/time to minimal volume) | 3 and 6 months
MVO2 max | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GAndre Ng, MB ChB, PhD, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester HNS trust, Leicester, England, United Kingdom